CLINICAL TRIAL: NCT07074704
Title: Transcranial Alternating Current Stimulation (tACS) as an Augmentation Treatment for Negative Symptoms and Cognitive Deficits in Long-term Hospitalized Schizophrenia Patients
Brief Title: tACS to Improve Negative Symptoms & Cognition in Long-term Hospitalized Schizophrenia Patients.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Weiqing Liu, Dr., Tongji University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDJWWLZL
Record Dates: First submitted 2025-06-23; First posted 2025-07-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Negative Symptoms in Schizophrenia; Cognition Function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TACS sham stimulation group (Sham Comparator): The intervention lasted for 10 days, with tACS stimulation performed twice a day for 40 minutes each time, using a current of 0 mA.
  Interventions: Device: Sham Comparison
- tACS Real stimulation group (Experimental): The intervention lasted for 10 days, with tACS stimulation performed twice a day for 40 minutes each time, using a current of 15 mA.
  Interventions: Device: Hi-tACS

INTERVENTIONS:
Device: Hi-tACS — Sham tACS intervention (0 mA) Twice a day, 40 min each time, for 10 days tACS intervention (15 mA) Twice a day, 40 minutes each time, for 10 days
  Arms: tACS Real stimulation group
Device: Sham Comparison — Sham tACS intervention (0 mA) Twice a day, 40 min each time, for 10 days tACS intervention (15 mA) Twice a day, 40 minutes each time, for 10 days
  Arms: TACS sham stimulation group

SUMMARY:
This study aims to evaluate the efficacy of transcranial alternating current stimulation (tACS) on negative symptoms and cognitive function in long-term hospitalized patients with schizophrenia. At the same time, this study will explore the potential impact of relevant biomarkers and genetic factors on the efficacy of tACS intervention.

DETAILED DESCRIPTION:
1. Research purpose (1) This study aims to explore the synergistic therapeutic effect of tACS on negative symptoms and cognitive function in long-term hospitalized schizophrenia patients; (2) Using emotion-induced EEG activity in a virtual reality context as a biomarker, analyze its correlation with the clinical efficacy of tACS.
2. Expected results (1) It is confirmed that tACS can improve negative symptoms and cognitive function in long-term hospitalized schizophrenia patients; (2) Biomarkers can be used to predict the efficacy of tACS in improving negative symptoms and cognitive function in long-term hospitalized schizophrenia patients, and guide clinical precision application.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for long-term hospitalized schizophrenia patients:

  1. Diagnosed with DSM-5 schizophrenia and hospitalized for more than half a year
  2. Aged between 18 and 65 years old
  3. Willing to participate in the study and sign the informed consent
  4. Stable condition, PANSS total score changed less than 15% at least 2 months before the study.
  5. Education level above primary school
  6. Normal vision or normal after correction

Inclusion criteria for normal control group:

1. No diagnosed mental illness
2. Aged between 18 and 65 years old
3. Willing to participate in the study and sign the informed consent
4. Education level above primary school
5. Normal vision or normal after correction
6. Residents living in Pudong community

Exclusion Criteria:

Exclusion criteria for long-term hospitalization of schizophrenia patients:

1. Combined diagnosis of other mental illnesses in DSM-5
2. History of severe neurological diseases, epilepsy, craniocerebral trauma, etc.
3. Severe organic diseases of the heart, liver, kidney and other organs that are unstable
4. Infectious skin diseases
5. Use of other drugs that affect the results during the study, such as benzodiazepines, non-benzodiazepine sedatives, and psychostimulants
6. Pregnant or lactating women
7. Patients with claustrophobia
8. Patients with alcohol, drugs Abuse history
9. Patients who have received TACS treatment in the past and have no effect or intolerance

Exclusion criteria for normal control group:

1. Patients with a history of severe neurological diseases, epilepsy, craniocerebral trauma, etc.
2. Patients with severe organic diseases that cause instability of organs such as heart, liver, and kidney
3. Patients with infectious skin diseases
4. During the study, drugs that affect the results were used in combination, such as benzodiazepines, non-benzodiazepine sedatives, and psychostimulants
5. Pregnant or lactating women
6. Patients with claustrophobia
7. Patients with a history of alcohol and drug abuse -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Eye Tracking | Day 1 before tACS intervention
  Binocular saccade amplitude and direction
Eye Tracking | Day 1 after tACS intervention
  Binocular saccade amplitude and direction
EEG | Day 1 before tACS intervention
  resting EEG power spectrum
EEG | Day 1 after tACS intervention
  resting EEG power spectrum
Brief Negative Symptom Scale (Bnss) | Day 1 before tACS intervention
  The Brief Negative Symptom Scale (BNSS) ranges from 0 to 78, with higher scores indicating more severe negative symptoms.
Brief Negative Symptom Scale (Bnss) | Day 4 after tACS intervention
  The Brief Negative Symptom Scale (BNSS) ranges from 0 to 78, with higher scores indicating more severe negative symptoms.
MATRICS Consensus Cognitive Battery，MCCB | Day 1 before tACS intervention
  The MATRICS Consensus Cognitive Battery (MCCB) does not have a fixed total score range, as it consists of multiple tests assessing different cognitive domains. Each domain score is standardized as a T-score, typically ranging from approximately 0 to 100, with higher scores indicating better cognitive performance.
MATRICS Consensus Cognitive Battery，MCCB | Day 4 after tACS intervention
  The MATRICS Consensus Cognitive Battery (MCCB) does not have a fixed total score range, as it consists of multiple tests assessing different cognitive domains. Each domain score is standardized as a T-score, typically ranging from approximately 0 to 100, with higher scores indicating better cognitive performance.
The Clinical Assessment Interview Scale | Day 1 before tACS intervention
  The Clinical Assessment Interview Scale for Negative Symptoms (CAINS) ranges from 0 to 52 , with higher scores indicating more severe negative symptoms.
The Clinical Assessment Interview Scale | Day 4 after tACS intervention
  The Clinical Assessment Interview Scale for Negative Symptoms (CAINS) ranges from 0 to 52 , with higher scores indicating more severe negative symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pudong New Area Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT07074704/Prot_000.pdf
  • Informed Consent Form (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT07074704/ICF_001.pdf